CLINICAL TRIAL: NCT04854213
Title: PRELUDE-1 (Prospective Evaluation of Radiotherapy-induced Biologic Effects in Colorectal Cancer Oligometastatic Patients with LUng-limited Disease: Evolution of Cancer Genetics and Regulatory Immune Cells)
Acronym: PRELUDE-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 88/20
Record Dates: First submitted 2021-04-09; First posted 2021-04-22 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer Metastatic
Keywords: SBRT; liquid biopsy; metastatic disease; cancer genetics; NGS; omCRC
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liquid biopsy (Other): Blood samples for liquid biopsy
  Interventions: Device: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Device: Stereotactic Body Radiation Therapy (SBRT) — Radiation treatment

SUMMARY:
PRELUDE-1 study is a pilot intervention trial that aims to describe the immunologic and genetic evolutions induced by stereotactic body radiationtherapy (SBRT) treatment in oligometastatic Colorectal Cancer (omCRC) patients with two-three nodules lung-limited disease.

DETAILED DESCRIPTION:
PRELUDE-1 study is a monocentric pilot interventional trial. The study concerns all patients enrolled with a diagnosis of oligometastatic Colorectal Cancer (omCRC) with two-three nodules lung-limited disease and treated with SBRT technique. SBRT will be delivered according to a risk-adapted protocol.

Tumor genetic background will be assessed on primary FFPE (Formalin Fixed Paraffin Embedded) tissues. Liquid biopsy will be done on blood samples collected before radiotherapy (RT) start and after 40 days to monitor tumor DNA evolution. The most direct method to assess cancer genetics relies on sampling of tumor DNA and its characterization through whole genome sequencing techniques (NGS, Next Generation Sequencing).

The study will last 48 months, divides as follow: 24 months of enrollment phase and up to 24 months of follow-up. Follow-up will be performed on the 40th day after the end of radiation treatment and then every 3 months until progression.

ELIGIBILITY:
Inclusion Criteria:

* Age <80 years
* Cytological or histological diagnosis of colorectal adenocarcinoma
* Two or three asymptomatic lung nodules smaller than 25 mm
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Available Formalin Fixed Paraffin Embedded (FFPE) of resected primary tumor
* Negative pregnancy test for all potentially childbearing women
* Patient candidates to SBRT

Exclusion Criteria:

* Previous systemic anti-tumor treatments (allowed treatment with capecitabine or fluorouracil and radiotherapy in the neoadjuvant setting of rectal tumors with therapy terminated at least 6 months before)
* Neutrophils <2000/mm³ or platelets <100.000/mm³ or hemoglobin <9 g/dl; serum creatinine level> 1.5 times the maximum normal value; GOT and/or GPT >5 times the maximum normal value and/or bilirubin level >3 times the maximum normal value
* Previous or concomitant malignant neoplasms (excluding basal or spinocellular cutaneous carcinoma or in situ carcinoma of the uterine cervix)
* Active or uncontrolled infections
* Other concomitant uncontrolled diseases or conditions contraindicating the study drugs at clinician evaluation
* Presence of brain metastases
* Refusal or inability to provide informed consent
* Impossibility to guarantee follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of SBRT in inducing a regressive genetic trajectory of KRAS gene (evaluated by NGS technique) after SBRT treatment. | 40 days after the end of RT
  A genetic regressive trajectory is defined as KRAS mutated (any mutation) before SBRT and wild-type after SBRT (mutKRAS before SBRT→wtKRAS after SBRT). The sample size of the study is planned on this genetic trajectory, assuming a frequency of the phenomenon of 1/130 (as desumed from literature review). To be exhaustive, other realistic combinations are: wtKRAS→wtKRAS; mutKRAS→mutKRAS; wtKRAS→mutKRAS. Other assumptions for sample size calculation are: an alpha value of 0.05; a priori successful events rate of 0.077; 1-beta=0.60.

SECONDARY OUTCOMES:
To evaluate the response according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria, version 1.1 including any eventual abscopal effect. | Up to 24 months after the end of RT
To evaluate the responses' duration (measured from the time of documented objective response until documented tumor progression). | Up to 24 months after the end of RT
To evaluate the progression-free (PFS) survival (from the data of treatment start untill progression). | Up to 24 months after the end of RT
The toxicity, which will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) of the National Cancer Institute, version 5.0, November 27, 2017. | Up to 24 months after the end of RT
  The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline. Higher scores mean worse outcome.
Tumor immune microenvironment in primary tumour | 40 days after the end of RT
  Evaluate the tumor immune microenvironment (in particular the number of CD3+/CD8+/Granzyme B+ lymphocytes) of primary CRCs by immunohistochemistry (IHC).
Metabolic response (exploratory studies) | 40 days after the end of RT
  Assess the value of metabolic response by FDG-PET (fluorodeoxyglucose positron emission tomography) through SUV (Standardized Uptake Value) percentage modifications [(SUV after SBRT-SUV before SBRT/SUV before SBRT)x100].

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Muto, MD, Principal Investigator — National Cancer Institute of Naples; Alessandro Ottaiano, MD, Principal Investigator — National Cancer Institute of Naples
Locations (1):
- Istituto Nazionale Tumori - Fondazione G. Pascale, Napoli, NAPOLI, Italy